CLINICAL TRIAL: NCT05024747
Title: A Randomized, Open Label, Single Center, Single Dose, Two Period, Two Sequence Crossover Bioequivalence Study of 21 mg Nicotine Transdermal Patches (NicoDerm CQ, GSK Dungarvan) Compared to the Current Marketed 21 mg Nicotine Transdermal Patches (NicoDerm CQ, Alza) in Healthy Adult Smokers
Brief Title: A Bioequivalence Study of 21 Milligram (mg) Nicotine Transdermal Patches (NicoDerm CQ, GlaxoSmithKline [GSK] Dungarvan) Compared to the Current Marketed 21 mg Nicotine Transdermal Patches (NicoDerm CQ, Alza) in Healthy Adult Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 217756
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Product (Experimental): Participants will receive a single NicoDerm CQ patch (GSK Dungarvan) placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours.
  Interventions: Drug: NicoDerm CQ patch (GSK Dungarvan)
- Reference Product (Active Comparator): Participants will receive a single NicoDerm CQ patch (Alza) placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours.
  Interventions: Drug: NicoDerm CQ (Alza)

INTERVENTIONS:
Drug: NicoDerm CQ patch (GSK Dungarvan) — A single patch of a NicoDerm CQ (GSK Dungarvan) 21 mg per system of 22 centimeter square (cm^2) surface area will be placed topically.
  Arms: Test Product
Drug: NicoDerm CQ (Alza) — A single patch of a NicoDerm CQ (Alza) 21 mg/system of 22 cm^2 surface area will be placed topically.
  Arms: Reference Product

SUMMARY:
The purpose of this study is to assess the bioequivalence of the 21mg nicotine transdermal patch from GSK Dungarvan (Test) compared to the 21mg nicotine transdermal patch currently manufactured by Alza (Reference).

DETAILED DESCRIPTION:
This is a 2-arm, single center, single dose, open-label, randomized, two-sequence, two-period crossover, bioequivalence study in healthy adult smokers that have smoked more than 10 cigarettes per day for 1 year prior to initial dose. Carry-over effects will be avoided by a wash-out interval of at least 2 days (but no more than 4 days) from patch removal in the first treatment period to subsequent patch application. The study will consist of an ambulant screening day within 21 days prior first patch application.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, as determined by medical evaluation, including a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead Electrocardiogram (ECG) or clinical laboratory tests.
* Body Mass Index (BMI) of 19 to 27 kilogram/meter Squared (kg/m^2); and a total body weight >50 kg (110 Pound-Mass [lbs]).
* Any female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 5 days after the last dose of assigned treatment. Female participant who are not of childbearing potential must meet requirements of protocol.
* Participants admits to having smoked more than 10 cigarettes per day for the preceding one year (prior to initial dose).
* Participant with two negative tests (one at screening and one at check in Day-2) for active COVID-19, separated by > 24 hours.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK Consumer Health (CH) employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving any investigational product(s) within 30 days before first dosing.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A Participant who is pregnant as confirmed by a positive serum pregnancy test or intending to become pregnant over the duration of the study.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients ethylene vinyl acetatecopolymer, polyisobutylene and high density polyethylene.
* Diagnosis of long QT syndrome or corrected QT (QTc) > 450 Millisecond (msec) for a male participant and > 470 msec for a female participant at screening.
* A participant unwilling or unable to comply with Lifestyle Considerations described in this protocol.
* Participant is unwilling to abstain from tobacco or nicotine-containing product use during the study (from check-in to the completion of the last pharmacokinetics (PK) blood sampling). Expired carbon monoxide (CO) measurement immediately prior to randomization (first treatment session) and dosing (second treatment session) should be less than or equal to (<=) 10 parts per million (ppm) for the participant to be dosed.
* Participant has used chewing tobacco, tobacco products or electronic cigarettes other than cigarettes within 21 days of Visit 1.
* Use of any medication (including over-the-counter medications and herbal remedies) within 2 weeks before first scheduled study drug administration or within < 10 times the elimination half-life of the respective drug (whichever is longer), or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:

  • systemic contraceptives and hormone replacement therapy, as long as female participant is on stable treatment for at least 3 months and continues treatment throughout the study.
* Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation, as assessed by the Investigator or medically qualified designee.
* A participant with a positive urine drug screen, for Tetrahydrocannabinol (THC), amphetamine, cocaine, 3,4-methylenedioxy-N-methylamphetamine (MDMA)/ecstasy, methamphetamine, or opiates.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
* participant with signs and symptoms suggestive of COVID-19 (i.e. fever, cough, etc) within 14 days of inpatient admission.
* Participant with known COVID-19 positive contacts in the past 14 days.
* Presence of tattoo, excessive hair (including shaved hair) or scarring on the test site on the back which in the opinion of the investigator would interfere with the study assessments.
* Participant who currently in the opinion of the investigator, after medical review, has any of the following conditions:

  * Thrombophlebitis, thromboembolic disorders
  * A history of deep vein thrombophlebitis or thromboembolic disorders
  * Cerebrovascular or coronary artery disease (current or history)
  * Valvular heart disease with complications
  * Severe hypertension
  * Diabetes with vascular involvement
  * Headaches with focal neurological symptoms
  * Major surgery with prolonged immobilization.
* Surgical procedures or use of topical pharmacologic treatments directly over the test site(s) within 90 days before enrollment.
* A participant with any condition possibly affecting drug absorption, distribution, metabolism or excretion of any drug substance but not limited to any of the following:

  * History or current evidence of dermatologic disorders/skin diseases including sunburn and keloids, that may interfere with the transdermal absorption of the study drug(s) at the test site;
  * History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (>=1.4 milligram per deciliter [mg/dL]) or Blood urea nitrogen (BUN) (>=25 mg/dL) or the presence of clinically significant abnormal urinary constituents (e.g.

albuminuria);

* History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A candidate will be excluded if more than one of the following lab value deviations are found: 1) Aspartate transaminase/Serum glutamic oxaloacetic transaminase (AST/SGOT) (>= 1.2 upper limit of normal [ULN]), Alanine transaminase/Serum glutamic pyruvic transaminase (ALT/SGPT) (>= 1.2 ULN), 2) Gamma glutamyl transpeptidase (GGT) (>= 1.2 ULN), Alkaline phosphatase (ALP) (>= 1.2 ULN), 3) bilirubin (>= 1.0 mg/dL) or Creatine kinase (CK) (>= 3 to 5 ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the Investigator;
* Evidence of urinary obstruction or difficulty in voiding at screening.

  * Evidence, as reported by an alcohol breath testing during screening, for current alcohol abuse or reports a regular average alcohol consumption exceeding 18 gram (g) (women) or 35 g (men) of pure alcohol per day, i.e., 1 drink/day for women or 2 drinks/day for men (1 drink = 5 ounce (oz) of wine or 12 oz of beer or 1.5 oz of hard liquor) within 6 months of screening.
  * participant reported regular consumption of > 5 cups of coffee or tea per day (or equivalent consumption of >= 500 mg xanthine per day using other products).
  * Participant reports consumption of any drug metabolizing enzyme (e.g., CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (e.g., broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort etc.) within 2 weeks prior to dosing.
  * Positive results at screening in any of the virology tests for human immunodeficiency virus-Ab (HIV-ab), hepatitis C virus-Ab (HCV-Ab), Hepatitis B surface antigen (HBsAg) and Hepatitis B Core Antibody (HBc-Ab) (Immunoglobulin G [IgG] + Immunoglobulin M [IgM]).
  * Performance of unaccustomed strenuous physical exercise (body building, high performance sports) from 2 weeks prior to dosing.
  * Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the Investigator's opinion may pose a risk to the candidate.
  * A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
  * Participation in a clinical trial with at least 470ml blood drawn, or blood donation within 30 days prior to the start of the study.
  * Hemoglobin value <11.0 g/dL
  * Participants who have previously been enrolled in this study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK ClinicalTrials, Study Director
Locations (1):
- GSK Investigational Site, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United States from 01 September 2021 to 25 October 2021. A total of 22 participants were enrolled, out of which 21 participants were randomized and received treatment during two treatment periods.
Pre-assignment Details: Eligible participants received either NicoDerm CQ patch (GSK Dungarvan) Test or NicoDerm CQ (Alza) Reference for a total duration of 24 hours on Day 1 (Period 1) and Day 5 (Period 2). Same participants had multiple movement within the arms of two sequence levels (Test and reference). So, overall participant data was planned, analyzed and reported to avoid double-counting in disposition and baseline characteristics.
Groups:
- NicoDerm CQ Dungarvan First, Then NicoDerm CQ Alza: Participants received a single-dose of 21 milligrams (mg) of NicoDerm CQ patch (GSK Dungarvan) Test on Day 1 (Period 1) and NicoDerm CQ (Alza) Reference on Day 5 (Period 2) placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours. Two periods were separated by 24 hours wash-out. The patch that was applied during Period 2 was not applied to the same position as the patch that was applied during Period 1 but on the upper back of the contralateral side of the body.
- NicoDerm CQ Alza First, Then NicoDerm CQ Dungarvan: Participants received a single-dose of 21 mg of NicoDerm CQ (Alza) Reference on Day 1 (Period 1) and NicoDerm CQ patch (GSK Dungarvan) Test on Day 5 (Period 2) placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours. Two periods were separated by 24 hours wash-out. The patch that was applied during Period 2 was not applied to the same position as the patch that was applied during Period 1 but on the upper back of the contralateral side of the body.
Period: Period 1 (Day 1 to 2)
Arm/Group | NicoDerm CQ Dungarvan First, Then NicoDerm CQ Alza | NicoDerm CQ Alza First, Then NicoDerm CQ Dungarvan
Started | 11 | 10
Completed | 10 | 5
Not Completed | 1 | 5
Not completed — Protocol Violation | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Patch fall off or patch is inadvertently removed by the participant | 0 | 1
Period: Wash-out (Day 3)
Arm/Group | NicoDerm CQ Dungarvan First, Then NicoDerm CQ Alza | NicoDerm CQ Alza First, Then NicoDerm CQ Dungarvan
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0
Period: Period 2 (Day 4 to 6)
Arm/Group | NicoDerm CQ Dungarvan First, Then NicoDerm CQ Alza | NicoDerm CQ Alza First, Then NicoDerm CQ Dungarvan
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all randomized participants who received at least one dose of study medication.
Groups:
- All Study Participants: Participants received a single-dose of 21 mg of either NicoDerm CQ patch (GSK Dungarvan) Test or NicoDerm CQ (Alza) Reference placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours on Day 1 (Period 1) and Day 5 (Period 2). Two periods were separated by 24 hours wash-out. The patch that was applied during Period 2 was not applied to the same position as the patch that was applied during Period 1 but on the upper back of the contralateral side of the body.
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (8.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Nicotine Concentration (Cmax) of NicoDerm CQ Dungarvan (Test) Compared to NicoDerm CQ, Alza (Reference)
Description: Cmax was the highest observed plasma nicotine concentration of NicoDerm CQ Dungarvan (Test) compared to NicoDerm CQ, Alza (Reference) was reported. Blood samples were collected at indicated time points. Pharmacokinetic analysis of NicoDerm CQ Dungarvan (Test) compared to NicoDerm CQ, Alza (Reference) was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed effects model fit to the log-transformed pharmacokinetic (PK) variables, as the dependent variable, treatment, and period as fixed effects. Geometric mean and CV of the geometric mean was presented. Comparison data of Test vs Reference was reported based on the baseline adjusted data.in statistical analysis 1.
Time Frame: Pre-dose (within 1 hour before dosing), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 24, 25, 26, 27, 28, 30, 32, and 36 hours post-dose in each treatment period
Population: The PK population was defined as all randomized participants who completed both periods, and who had no major protocol deviations concerning PK regardless of patch adhesion score.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Groups:
- NicoDerm CQ Dungarvan (Test): Participants received a single dose of 21 mg of NicoDerm CQ patch (GSK Dungarvan) Test placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours either on Day 1 (Period 1) or Day 5 (Period 2). Two periods were separated by 24 hours wash-out. The patch that was applied during Period 2 was not applied to the same position as the patch that was applied during Period 1 but on the upper back of the contralateral side of the body.
- NicoDerm CQ Alza (Reference): Participants received a single dose of 21 mg of NicoDerm CQ (Alza) Reference placed topically under fasted conditions to the upper part of the back for a total duration of 24 hours either on either (Period 1) or Day 5 (Period 2). Two periods were separated by 24 hours wash-out. The patch that was applied during Period 2 was not applied to the same position as the patch that was applied during Period 1 but on the upper back of the contralateral side of the body.
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 15 | 15
Nanograms per milliliter (ng/mL) | 23.554 (20.3) | 24.478 (22.9)
Statistical Analysis 1: Comparison: NicoDerm CQ Dungarvan (Test) vs NicoDerm CQ Alza (Reference); Statistical comparison was analyzed between Test vs Reference based on Baseline Adjusted Data; Test type: Other; Ratio T/R = 96.68, 90% CI 2-sided [90.00 to 103.85]

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to Time t (AUC [0-t]) of NicoDerm CQ Dungarvan (Test) Compared to NicoDerm CQ, Alza (Reference)
Description: Area under the plasma concentration versus time curve from time zero to time t, where t was the time of the last measurable plasma concentration of nicotine, estimated, computed using the linear trapezoidal rule. Blood samples were collected at indicated time points. Pharmacokinetic analysis of NicoDerm CQ Dungarvan (Test) compared to NicoDerm CQ, Alza (Reference) was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed effects model fit to the log-transformed PK variable, as the dependent variable, treatment, and period as fixed effects. Geometric mean and CV of the geometric mean was presented. Comparison data of Test vs Reference was reported based on the baseline adjusted data.in statistical analysis 1.
Time Frame: Pre-dose (within 1 hour before dosing), 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 24, 25, 26, 27, 28, 30, 32, and 36 hours post-dose
Population: Analysis was performed using PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram per milliliter (h*ng/mL)
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 15 | 15
Hour*nanogram per milliliter (h*ng/mL) | 529.464 (24.6) | 564.085 (23.4)
Statistical Analysis 1: Comparison: NicoDerm CQ Dungarvan (Test) vs NicoDerm CQ Alza (Reference); Statistical comparison was analyzed between Test vs Reference based on Baseline Adjusted Data; Test type: Other; Ratio T/R = 92.37, 90% CI 2-sided [85.45 to 99.84]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated From Time Zero to Infinity (AUC [(0-inf]) of NicoDerm CQ Dungarvan (Test) Compared to NicoDerm CQ, Alza (Reference)
Description: Area under the plasma concentration versus time curve calculated from time zero to infinity. AUC0-inf = AUC0-t + C(t)/λz. C(t)- Concentration at the last measurable sampling time point and λz- terminal elimination rate constant. Blood samples were collected at indicated time points. Pharmacokinetic analysis of NicoDerm CQ Dungarvan (Test) compared to NicoDerm CQ, Alza (Reference) was conducted using standard non-compartmental analysis. Analysis was performed using a linear mixed effects model fit to the log-transformed PK variable, as the dependent variable, treatment, and period as fixed effects. Geometric mean and CV of the geometric mean was presented. Comparison data of Test vs Reference was reported based on the baseline adjusted data.in statistical analysis 1.
Time Frame: as for outcome 2
Population: Analysis was performed using PK population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 15 | 15
h*ng/mL | 537.518 (24.9) | 571.211 (24.0)
Statistical Analysis 1: Comparison: NicoDerm CQ Dungarvan (Test) vs NicoDerm CQ Alza (Reference); Statistical comparison was analyzed between Test vs Reference based on Baseline Adjusted Data; Test type: Other; Ratio T/R = 92.54, 90% CI 2-sided [85.63 to 100.01]

4. Secondary Outcome: Terminal Elimination Rate Constant (Lambda z) of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) of Patches
Description: Terminal elimination rate constant for plasma nicotine computed as the slope of the regression line of ln (C(t)) on time. The regression should generally involve at least 3 consecutive measurable concentrations that decrease over time. Blood samples were collected at indicated time points. Pharmacokinetic analysis of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 2
Population: Analysis was performed using PK population.
Measure: Median (Inter-Quartile Range); unit: Per hour
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 15 | 15
Per hour | 0.2141 [0.18266 to 0.23855] | 0.2475 [0.19543 to 0.26550]
Statistical Analysis 1: Comparison: NicoDerm CQ Dungarvan (Test) vs NicoDerm CQ Alza (Reference); Statistical comparison was analyzed between Test vs Reference; Test type: Other; p = 0.0833, Wilcoxon Signed Rank Test; Hodges- Lehmann's median difference = -0.0192, 95% CI 2-sided [-0.0542 to 0.0044]

5. Secondary Outcome: Maximum Plasma Nicotine Concentration (Tmax) of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) Patches
Description: Time to maximum plasma nicotine concentration of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) patches was reported. Blood samples were collected at indicated time points. Pharmacokinetic analysis of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) patches was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 2
Population: Analysis was performed using PK population.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 15 | 15
Hours | 4.000 [3.0000 to 10.0000] | 18.000 [4.0000 to 18.0000]
Statistical Analysis 1: Comparison: NicoDerm CQ Dungarvan (Test) vs NicoDerm CQ Alza (Reference); Statistical comparison was analyzed between Test vs Reference; Test type: Other; p = 0.0205, Wilcoxon Signed Rank Test; Hodges- Lehmann's median difference = -6.0000, 95% CI 2-sided [-10.5000 to 0.0000]

6. Secondary Outcome: Elimination Half-Life (t1/2) of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) Patches
Description: t1/2 was apparent elimination half-life. The elimination half-life computed as t1/2 = ln(2)/ λz). Blood samples were collected at indicated time points. Pharmacokinetic analysis of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) patches was conducted using standard non-compartmental analysis.
Time Frame: as for outcome 2
Population: Analysis was performed using PK population.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 15 | 15
Hours | 3.2376 [2.90566 to 3.79479] | 2.8001 [2.61074 to 3.54677]
Statistical Analysis 1: Comparison: NicoDerm CQ Dungarvan (Test) vs NicoDerm CQ Alza (Reference); Statistical comparison was analyzed between Test vs Reference; Test type: Other; p = 0.0946, Wilcoxon Signed Rank Test; Hodges- Lehmann's median difference = 0.3225, 95% CI 2-sided [-0.0949 to 0.6810]

7. Secondary Outcome: Number of Participants With Adhesion Score of NicoDerm CQ Dungarvan (Test) and NicoDerm CQ, Alza (Reference) Patches
Description: Adhesion to skin assessed by FDA recommended 0-4 scoring system. The scoring for adhesion of patches was indicated as follows: Score 0 ( Greater than or equal to [>=] 90% Adhered [essentially no lift off the skin]), Score 1 (>= 75% to less than [<] 90% Adhered [some edges only lifting off the skin]), Score 2 (>= 50% to < 75% Adhered [less than half of the patch lifting off the skin]), Score 3 (greater than [>] 0% to < 50% Adhered but not detached [more than half of the patch lifting off the skin without falling off]), and Score 4 (0% adhered [patched completely detached]).
Time Frame: At 0, 6, 12, 18 and 24 hours post-dose
Population: Analysis was performed using safety population. Out of 21 participants, 16 participants who were dosed with NicoDerm CQ Dungarvan (Test) and 20 participants dosed with NicoDerm CQ Alza (Reference).
Measure: Count of Participants; unit: Participants
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 16 | 20
Participants
  0 hour (Immediately After Patch Application): At Score 0 | 16 | 20
  0 hour (Immediately After Patch Application): At Score 1 | 0 | 0
  0 hour (Immediately After Patch Application): At Score 2 | 0 | 0
  0 hour (Immediately After Patch Application): At Score 3 | 0 | 0
  0 hour (Immediately After Patch Application): At Score 4 | 0 | 0
  6 Hours After Patch Application: At Score 0 | 11 | 14
  6 Hours After Patch Application: At Score 1 | 5 | 6
  6 Hours After Patch Application: At Score 2 | 0 | 0
  6 Hours After Patch Application: At Score 3 | 0 | 0
  6 Hours After Patch Application: At Score 4 | 0 | 0
  12 Hours After Patch Application: At Score 0 | 5 | 10
  12 Hours After Patch Application: At Score 1 | 11 | 10
  12 Hours After Patch Application: At Score 2 | 0 | 0
  12 Hours After Patch Application: At Score 3 | 0 | 0
  12 Hours After Patch Application: At Score 4 | 0 | 0
  18 Hours After Patch Application: At Score 0 | 4 | 6
  18 Hours After Patch Application: At Score 1 | 12 | 13
  18 Hours After Patch Application: At Score 2 | 0 | 0
  18 Hours After Patch Application: At Score 3 | 0 | 1
  18 Hours After Patch Application: At Score 4 | 0 | 0
  24 Hours After Patch Application: At Score 0 | 2 | 5
  24 Hours After Patch Application: At Score 1 | 14 | 14
  24 Hours After Patch Application: At Score 2 | 0 | 0
  24 Hours After Patch Application: At Score 3 | 0 | 0
  24 Hours After Patch Application: At Score 4 | 0 | 1

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs (TEAEs)
Description: TEAEs were defined as any adverse events (AEs) that first occurred on or after the date and time of patch administration. Any AE that first occurred pre-dose but worsened in severity after the first patch administration was also considered a TEAE. An SAE was any untoward medical occurrence that at any dose met one, more of the following criteria: results in death, life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent, significant disability/incapacity, a congenital abnormality/birth defect, an important medical event. A TEAE was any event emerging or manifesting at or after the initiation of treatment with an IP or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the IP or medicinal product. Number of Participants with TEAEs and serious TEAEs were reported.
Time Frame: From start of study drug administration up to end of study visit (up to Day 6)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
Number analyzed (Participants) | 16 | 20
Participants
  Participants with TEAEs | 7 | 11
  Participants with Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to end of study visit (up to Day 6)
Description: Analysis was performed using safety population. Out of 21 participants, 16 participants who were dosed with NicoDerm CQ Dungarvan (Test) and 20 participants dosed with NicoDerm CQ Alza (Reference).
Arm/Group | NicoDerm CQ Dungarvan (Test) | NicoDerm CQ Alza (Reference)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 7/16 | 11/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NicoDerm CQ Dungarvan (Test) (N=16) | NicoDerm CQ Alza (Reference) (N=20)
Dizziness (Nervous system disorders) | 2 (4) | 4 (5)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 6 (6) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematocrit increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Red blood cell count increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT05024747/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT05024747/SAP_001.pdf